CLINICAL TRIAL: NCT02911571
Title: Prospective Multicenter Study to Measure the Impact of MMprofiler on Treatment Intention in Active Multiple Myeloma Patients
Brief Title: PRospective Multiple Myeloma Impact Study
Acronym: PROMMIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SkylineDx (Industry)
Collaborators: Medex15 (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROMMIS
Record Dates: First submitted 2016-09-15; First posted 2016-09-22 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MMprofiler SKY92 (Experimental): Eligible patients will have their bone marrow biopsy sample analyzed for the prognostic MMprofiler SKY92 gene signature
  Interventions: Device: MMprofiler SKY92 gene signature

INTERVENTIONS:
Device: MMprofiler SKY92 gene signature — MMprofiler is a gene expression assay system for detection of the presence (or absence) of the SKY92 "high-risk" gene signature to aid in the determination of the Multiple Myeloma patient's prognosis

SUMMARY:
This will be a prospective, case-only, study to measure the impact of MMprofiler on treatment intention decisions in Multiple Myeloma patients.

DETAILED DESCRIPTION:
This will be a prospective, case-only, study to measure the impact of MMprofiler on treatment intention decisions in MM patients.

Eligible patients will have their tumor sample analyzed for the prognostic MMprofiler SKY92, several cytogenetic markers, gene expression markers, and gene expression clusters.

A total of 250 patients will be enrolled from up to 9 US centers. Patients will be followed 5 years after diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Potentially multiple myeloma according to IMWG criteria
* Candidates for systemic treatment

Exclusion Criteria:

* ECOG Performance Status > 3
* Tumor sample that fails QA or QC criteria for MMprofiler

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in treatment intention | Treatment intention is measured before MMprofiler SKY92 and within 4 weeks after MMprofiler
  Change in treatment intention will be assessed with a physician questionnaire pre- and post MMprofiler assessment

SECONDARY OUTCOMES:
3 year Progression Free Survival | 3 years after diagnosis
  Duration from start of the treatment to disease progression or death (regardless of cause of death), whichever comes first.
3 year Overall Survival | 3 years after diagnosis
  Duration from start of the treatment to death (regardless of cause of death).
5 year Progression Free Survival | 5 years after diagnosis
  Duration from start of the treatment to disease progression or death (regardless of cause of death), whichever comes first.
5 year Overall Survival | 5 years after diagnosis
  Duration from start of the treatment to disease progression or death (regardless of cause of death), whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Saad Usmani, MD, Principal Investigator — Charlotte Mecklenburg Hospital Authority, Carolinas HealthCare System
Locations (9):
- United States (9):
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Medical Center,, Winston-Salem, North Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No